CLINICAL TRIAL: NCT03705013
Title: Observational Study of Sub-populations From "A Longitudinal Study of Cologuard in an Average Risk Population Assessing a Three Year Test Interval"/Protocol 2014-01 Post-Approval Study
Brief Title: Observational Study of Sub-populations From Cologuard Post-Approval Study (2014-01)
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-09
Record Dates: First submitted 2018-09-24; First posted 2018-10-15 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: Cologuard
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Baseline Cologuard positive and negative colonoscopy: Those whose Cologuard T0 result was positive and colonoscopy result was negative.
  Interventions: Other: Cologuard
- Baseline Cologuard positive and no colonoscopy: Those whose Cologuard T0 result was positive and subject declined to complete a colonoscopy per protocol.
  Interventions: Other: Cologuard
- 3-year follow-up Cologuard positive and negative colonoscopy: Those whose Cologuard result at T3 was positive and colonoscopy result at T3 was negative.
  Interventions: Other: Cologuard
- 3-year follow-up Cologuard positive and no colonoscopy: Those whose Cologuard result at T3 was positive and subject declined to complete a colonoscopy per protocol.
  Interventions: Other: Cologuard

INTERVENTIONS:
Other: Cologuard — Observational

SUMMARY:
The primary endpoint is to obtain longitudinal information on four sub-populations from the Cologuard Post-Approval Study.

DETAILED DESCRIPTION:
Subjects who consented to enroll in Exact Sciences Protocol 2014-01, that fit one of the following sub-populations, will be asked to participate in the sub-study. Population 1 includes those whose Cologuard T0 result was positive and colonoscopy result was negative. Population 2 includes those whose Cologuard T0 result was positive and subject declined to complete a colonoscopy per protocol. Population 3 includes those whose Cologuard result at T3 was positive and colonoscopy result at T3 was negative. Population 4 includes those whose Cologuard result at T3 was positive and subject declined to complete a colonoscopy per protocol. Subjects that enrolled in the Exact Sciences Protocol 2014-01, who provided written informed consent to participate in this sub-study, will asked to complete the Follow-Up Questionnaire during a phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Subject falls into one of the 4 sub-populations
* Willing to provide informed consent

Exclusion Criteria:

* Death
* Investigator/sponsor decision
* Subject withdrew consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are four sub-populations of the Cologuard Post-Approval Study (2014-01) under observation: positive first Cologuard test and negative colonoscopy or no colonoscopy and positive 3-year follow-up Cologuard test and negative colonoscopy or no colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2019-11-16 (Actual)

PRIMARY OUTCOMES:
The number of subjects with discordant results that can be attributed to intercurrent disease | 3 years after positive Cologuard result
  A medical chart review and phone interview will be conducted for each subject. The Follow-Up Questionnaire will be completed during the phone interview.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Thomas C Lenzmeier, M.D., P.C., Glendale, Arizona
  - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - Cassidy Medical Group, Carlsbad, California
  - John D. Homan, MD, Newport Beach, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Innovative Research of West Florida, Clearwater, Florida
  - Homestead Medical Research, Homestead, Florida
  - Health Awareness Inc., Jupiter, Jupiter, Florida
  - Health Awareness Inc., Port St. Lucie, Port Saint Lucie, Florida
  - The Kaufmann Clinic, Atlanta, Georgia
  - Indiana University, Eskanazi Hospital, Regenstrief Health Center, Indianapolis, Indiana
  - Centennial Medical Group, Elkridge, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Nevada Family Care, Henderson, Nevada
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Family Practice Center of Wooster, Massillon, Ohio
  - Austin Regional Clinic, Austin, Texas
  - PCP for Life, Montgomery, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No